CLINICAL TRIAL: NCT02419508
Title: Additive Effect of Twice Daily Brinzolamide 1%/Brimonidine 0.2% Fixed Dose Combination as an Adjunctive Therapy to a Prostaglandin Analogue
Brief Title: SIMBRINZA® Suspension BID as an Adjunctive to Prostaglandin Analogue (PGA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLH694-P001; 2015-000736-15 (EudraCT Number); REec-2015-1723 (Registry Identifier: Registro Espanol de Estudios Clinicos)
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate; Prostaglandins, Synthetic; Bimatoprost; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SIMBRINZA + PGA (Experimental): Brinzolamide 1%/brimonidine 0.2% tartrate ophthalmic suspension, 1 drop instilled 2 times per day in affected eye(s) (09:00 and 21:00) plus designated prostaglandin analogue, 1 drop instilled in each eye once per day in the evening for 42 days
  Interventions: Drug: Brinzolamide 1%/brimonidine 0.2% tartrate ophthalmic suspension; Drug: Prostaglandin analogue
- Vehicle + PGA (Other): Brinz/brim vehicle, 1 drop instilled 2 times per day in affected eye(s) (09:00 and 21:00) plus designated prostaglandin analogue, 1 drop instilled in each eye once per day in the evening for 42 days
  Interventions: Drug: Brinz/brim vehicle; Drug: Prostaglandin analogue

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine 0.2% tartrate ophthalmic suspension
  Other Names: SIMBRINZA® suspension
  Arms: SIMBRINZA + PGA
Drug: Brinz/brim vehicle — Inactive ingredients used as a placebo for masking purposes
  Arms: Vehicle + PGA
Drug: Prostaglandin analogue
  Other Names: TRAVATAN® PQ (Travoprost ophthalmic solution with PQ, 0.004%); LUMIGAN® (Bimatoprost ophthalmic solution, 0.01%); XALATAN® (Latanoprost ophthalmic solution, 0.005%)

SUMMARY:
The purpose of this study is to evaluate the additive intraocular pressure (IOP) lowering effect of brinzolamide 1%/brimonidine 0.2% (dosed twice per day (BID)) when added to a prostaglandin analogue (PGA) in subjects with open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
This study consisted of 2 sequential phases: Screening/Eligibility Phase, followed by a Masked Treatment Phase (Phase II). Subjects were assigned into one of 3 PGA therapy groups for the duration of the study, based upon commercial availability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either open-angle glaucoma or ocular hypertension;
* Must sign an informed consent form;
* Mean IOP measurements at both the Eligibility 1 and 2 visits, in at least 1 eye (the same eye[s]) ≥ 19 and < 32 mmHg at 09:00.
* Willing and able to attend all study visits;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential who are pregnant, breast-feeding, intend to become pregnant during the study, or not using adequate birth control methods to prevent pregnancy throughout the study;
* Any form of glaucoma other than open-angle glaucoma or ocular hypertension;
* Ocular disease, trauma, infection, inflammation, pathology, or surgery as specified in the protocol;
* Any other conditions including severe illness which would make the subject, in the opinion of the Investigator, unsuitable for the study;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Ophtha, GCRA, Study Director — Alcon, a Novartis Company
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 37 sites located in Argentina (3), Australia (4), Canada (12), Chile (3), France (1), Germany (3), Greece (2), Israel (3), Spain (3), and United Kingdom (3).
Pre-assignment Details: Of the 290 subjects enrolled in the study, 102 were exited during the Screening/Eligibility period. This reporting group includes all randomized subjects. One randomized subject did not receive investigational product and is excluded from the Full Analysis Set and the Safety Analysis Set.
Period: Overall Study
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA
Started | 96 | 92
Full Analysis Set | 95 | 92
Safety Analysis Set | 95 | 92
Completed | 86 | 88
Not Completed | 10 | 4
Not completed — Adverse Event | 9 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other - Reason not specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who received a dose of study medication and had at least 1 of the 2 scheduled on-treatment visits [Full Analysis Set (FAS)].
Groups:
- Total: Total of all reporting groups
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA | Total
Number analyzed (Participants) | 95 | 92 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (10.70) | 67.9 (11.65) | 67.2 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 43 | 98
  Male | 40 | 49 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 29 | 52
  Not Hispanic or Latino | 72 | 62 | 134
  Unknown or Not Reported | 0 | 1 | 1
Baseline Diurnal IOP [Mean (Standard Deviation); unit: millimeters mercury (mmHg)] — IOP (fluid pressure inside the eye) was measured using Goldmann applanation tonometry and averaged over the 09:00 AM and 11:00 AM time points. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
  millimeters mercury (mmHg) | 22.8 (2.39) | 22.9 (2.32) | 22.8 (2.35)
Region of Enrollment [Count of Participants; unit: Participants]
  Europe, Australia | 45 | 44 | 89
  Latin America, Canada | 50 | 48 | 98

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (on PGA) in Diurnal IOP (Mean of 09:00 and 11:00 Time Points) at Week 6
Description: IOP (fluid pressure inside the eye) was measured using Goldmann applanation tonometry and averaged over the 09:00 AM and 11:00 AM time points. A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 6
Population: FAS. Only subjects with a value at both baseline and time point are included in the calculation of change.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA
Number analyzed (Participants) | 86 | 88
mmHg | -5.6 (2.72) | -2.1 (2.61)
Statistical Analysis 1: Comparison: SIMBRINZA + PGA vs Vehicle + PGA; Test type: Superiority; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: Mean Diurnal IOP at Week 6
Description: IOP (fluid pressure inside the eye) was measured using Goldmann applanation tonometry and averaged over the 09:00 AM and 11:00 AM time points. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye (study eye) contributed to the analysis.
Time Frame: Week 6
Population: FAS with data available
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA
Number analyzed (Participants) | 86 | 88
mmHg | 17.2 (3.49) | 20.9 (3.59)
Statistical Analysis 1: Comparison: SIMBRINZA + PGA vs Vehicle + PGA; Test type: Superiority; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: Mean Percentage Change From Baseline in Diurnal IOP at Week 6
Description: IOP (fluid pressure inside the eye) was measured using Goldmann applanation tonometry and averaged over the 09:00 AM and 11:00 AM time points. A more negative percent change from baseline indicates a greater improvement, i.e., a reduction of IOP. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 6
Population: FAS. Only subjects with a value at both baseline and time point are included in the calculation of change.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA
Number analyzed (Participants) | 86 | 88
percent change | -24.7 (12.17) | -9.5 (10.92)
Statistical Analysis 1: Comparison: SIMBRINZA + PGA vs Vehicle + PGA; Test type: Superiority; p < 0.001, Mixed Models Analysis

4. Secondary Outcome: Mean Change From Baseline in IOP at 11:00 at Week 6
Description: IOP (fluid pressure inside the eye) was measured using Goldmann applanation tonometry at 11:00 AM. A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 6
Population: FAS. Only subjects with a value at both baseline and time point are included in the calculation of change.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA
Number analyzed (Participants) | 95 | 92
mmHg
  Baseline | 22.4 (2.70) | 22.6 (2.69)
  Change from baseline: number analyzed (Participants) | 86 | 88
  Change from baseline | -7.0 (3.19) | -2.4 (2.78)
Statistical Analysis 1: Comparison: SIMBRINZA + PGA vs Vehicle + PGA; Test type: Superiority; p < 0.001, Mixed Models Analysis

5. Secondary Outcome: Mean Percentage Change From Baseline in IOP at 11:00 at Week 6
Description: IOP (fluid pressure inside the eye) was measured using Goldmann applanation tonometry at 11:00 AM. A more negative percent change from baseline indicates a greater improvement, i.e., a reduction of IOP. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 6
Population: FAS. Only subjects with a value at both baseline and time point are included in the calculation of change.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA
Number analyzed (Participants) | 86 | 88
percent change | -31.3 (14.81) | -10.8 (11.86)
Statistical Analysis 1: Comparison: SIMBRINZA + PGA vs Vehicle + PGA; Test type: Superiority; p < 0.001, Mixed Models Analysis

6. Secondary Outcome: Mean Change From Baseline in IOP at 09:00 at Week 6
Description: IOP (fluid pressure inside the eye) was measured using Goldmann applanation tonometry at 09:00 AM. Baseline is defined as the average of the 9:00 hour values at both Eligibility visits. A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 6
Population: FAS. Only subjects with a value at both baseline and time point are included in the calculation of change.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA
Number analyzed (Participants) | 95 | 92
mmHg
  Baseline | 23.4 (2.40) | 23.4 (2.22)
  Change from baseline: number analyzed (Participants) | 86 | 88
  Change from baseline | -4.9 (3.06) | -2.5 (2.87)
Statistical Analysis 1: Comparison: SIMBRINZA + PGA vs Vehicle + PGA; Test type: Superiority; p < 0.001, Mixed Models Analysis

7. Secondary Outcome: Mean Percentage Change From Baseline at 09:00 at Week 6
Description: IOP (fluid pressure inside the eye) was measured using Goldmann applanation tonometry at 9:00 AM. Baseline is defined as the average of the 9:00 hour values at both Eligibility visits.A more negative percent change from baseline indicates a greater improvement, i.e., a reduction of IOP. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 6
Population: FAS. Only subjects with a value at both baseline and time point are included in the calculation of change.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA
Number analyzed (Participants) | 86 | 88
percent change | -21.0 (13.36) | -10.9 (11.83)
Statistical Analysis 1: Comparison: SIMBRINZA + PGA vs Vehicle + PGA; Test type: Superiority; p < 0.001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Baseline through study completion, an average of 6 weeks.
Description: Adverse Events (AEs) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.This analysis population includes all subjects who received a dose of study medication (Safety Analysis Set).
Arm/Group | SIMBRINZA + PGA | Vehicle + PGA
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/92
Serious Adverse Events (participants affected / at risk) | 1/95 | 0/92
Other Adverse Events (participants affected / at risk) | 10/95 | 1/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIMBRINZA + PGA (N=95) | Vehicle + PGA (N=92)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIMBRINZA + PGA (N=95) | Vehicle + PGA (N=92)
Ocular hyperaemia (Eye disorders) | 5 (9) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT02419508/SAP_000.pdf
  • Study Protocol (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT02419508/Prot_001.pdf